CLINICAL TRIAL: NCT03622320
Title: Metabolic Syndrome in Early Onset Versus Late Onset Vitiligo
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Mogawer, Principal investigator, Cairo University
Other Study IDs: Vitiligo & Metabolic syndrome
Record Dates: First submitted 2018-07-16; First posted 2018-08-09 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2022-07

CONDITIONS: Metabolic Syndrome; Vitiligo
Keywords: insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Vitiligo; Insulin Resistance | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vitiligo patients: Vitiligo patients (100 NSV and 50 segmental) who will be further classified according to age of onset and blood sample will be taken
  Interventions: Other: Blood sample
- controls: Matching will be done taking into consideration age, sex, education and socio economic status, blood sample will be taken
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample for fasting blood sugar (FBS), High density lipoproteins (HDL), Triglycerides (TG) ,HOMA-IR, serum leptin

SUMMARY:
This study aims at detection of possible associated metabolic syndrome with vitiligo and assessment of possible contribution of the age of onset of vitiligo.

DETAILED DESCRIPTION:
This study aims at detection of incidence of metabolic syndrome in vitiligo patients and possible contribution of the age of onset of the disease. This involves detection of waist circumference, body mass index, index of central obesity, systolic and diastolic arterial blood pressure, fasting blood sugar, high density lipoproteins and triglycerides, in addition to insulin resistance as Homeostatic Model Assessment- insulin resisitance (HOMA-IR) and serum leptin in vitiligo patients. The outcomes will be correlated to extent/ severity/duration/ activity of vitiligo as well as to the age of onset. This is assumed to be of profound impact on vitiligo patients by properly assessing these patients for associated metabolic risk factors and helping prevent such metabolic derangements by detection of possible contributing factors such as insulin resistance and high serum adipokines as leptin.

Since there is temporal relation between nutrition, metabolic derangements and skin diseases where nutritional deficiencies as minerals, vitamins and fatty acids can lead to cutaneous manifestations and , on the other hand; skin diseases could contribute to metabolic derangements and nutritional deficiencies, the investigator's study will focus on nutrition and dietary habits and there possible contribution to any associated metabolic risk in vitiligo patients.

This is likely to open new horizons in the management of vitiligo, possibly through control of metabolic syndrome risk factors and insulin resistance as well as revealing possible temporal relation to dietary habits that are overlooked in vitiligo patients.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Patients with non-segmental vitiligo (NSV) and segmental vitiligo

Exclusion Criteria:

* Smoking
* Pregnancy
* Systemic steroid intake in the last 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Vitiligo patients presenting to Dermatology outpatient clinic (Kasr Alainy Teaching Hospitals, Cairo University).
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Central obesity as a Metabolic risk in vitiligo patients | one year
  Central obesity will be assessed using waist circumference in cm in vitiligo patients and control group as a risk factor for metabolic syndrome

SECONDARY OUTCOMES:
Arterial Blood Pressure as a Metabolic risk in vitiligo patients | one year
  Arterial Blood Pressure will be assessed in vitiligo patients and control group as a risk factor for metabolic syndrome
Fasting Blood pressure as a Metabolic risk in vitiligo patients | one year
  Fasting Blood pressure will be assessed in vitiligo patients and control group as a risk factor for metabolic syndrome
Serum Triglycerides and HDL | one year
  Serum Triglycerides and HDL will be assessed in vitiligo patients and control group as a risk factor for metabolic syndrome
Body mass index as a Metabolic risk in vitiligo patients | one year
  Body Mass index in kg/m2 will be assessed in vitiligo patients and control group as a risk factor for metabolic syndrome
Detection of insulin resistance in patients with vitiligo | one year
  This is via measuring HOMA-IR
Correlation between extent/ severity/duration/ activity of vitiligo and possible associated metabolic derangements. | one year
  This via detecting VASI, VES and VIDA scores for vitiligo patients
Correlation between extent/ severity/duration/ activity of vitiligo and the age of onset. | one year
  This via detecting VASI, VES and VIDA scores for vitiligo patients and relating to the age of onset
Detection of possible influence of dietary habits and its relation to metabolic derangements and disease progression | one year
  This via directly addressing dietary habits

CONTACTS AND LOCATIONS:
Overall Officials: Samar El-Tahlawi, MD, Principal Investigator — Cairo university, dermatology department
Locations (1):
- Cairo university hospitals, dermatology outpatient clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibrahim S, El-Tahlawi S, Mogawer RM, El Ansary M, Esmat S, El-Hawary M. Different vitiligo characteristics as predictors of increased risk of metabolic syndrome and insulin resistance: A case-control study. J Cosmet Dermatol. 2022 Dec;21(12):7170-7177. doi: 10.1111/jocd.15446. Epub 2022 Oct 25. PMID 36208004